CLINICAL TRIAL: NCT02939781
Title: Measuring Energy Expenditure Before and After Fever in Critically Ill Children
Brief Title: Measuring the Metabolic Cost of Fever
Acronym: IGUANA
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit to protocol
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 209010
Record Dates: First submitted 2016-10-11; First posted 2016-10-20 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2016-10

CONDITIONS: Child; Critical Illness; Fever
MeSH Terms: conditions — Critical Illness; Fever | interventions — Calorimetry, Indirect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Febrile critically ill children: Children above 10kg admitted to the paediatric intensive care unit at Great Ormond Street Hospital who are mechanically ventilated and have a high likelihood of developing a fever. Energy expenditure will be measured using indirect calorimetry at baseline, and continuously during fever, until fever subsides.
  Interventions: Device: Indirect calorimetry

INTERVENTIONS:
Device: Indirect calorimetry — Indirect calorimetry measurement at baseline (stable state), at onset of fever and continued till fever dehiscence

SUMMARY:
Fever is part of the body's immune response, often triggered by infection. Fever is commonly treated with medicines such as paracetamol, mainly because people feel unwell with fever. However fever does have a role in fighting infection: it enables the rest of the immune system to function more efficiently, and may directly stop bacteria and viruses from multiplying. In most cases however treating fever does not matter because the rest of the immune system can cope well enough to fight the infection (with or without additional treatment, like antibiotics).

In critically ill patients however any advantage in the fight against infection may be crucial. In a large observational study of adult patients in the intensive care unit, patients who developed an early fever with temperature between 38.5-39.5 degrees C fared relatively better than patients who were colder. So it is possible that in critical illness fever may be beneficial. However in critical illness the body does have limited energy resources. In order to raise the body temperature energy is required. However the investigators do not know how much energy is required to generate a fever in critically ill children. This study will aim to try and measure the energy required to generate a fever in a critically ill child. The investigators will measure energy expenditure directly in children admitted to the intensive care unit by measuring the levels of oxygen and carbon dioxide they breathe in and out (a method called indirect calorimetry). This will enable the investigators to judge whether the benefits of a fever can be justified by the energy costs in the energy depleted state that is critical illness.

ELIGIBILITY:
Inclusion Criteria:

- all children on the paediatric intensive care unit at Great Ormond Street Hospital who

1. are likely to or have developed a fever (suspected infection, following trauma, post major surgery)
2. are over 10kg (approx 1 year of age)
3. are invasively ventilated

Exclusion Criteria:

- Children who

1. have a brain injury, where active temperature control may be instituted
2. patients post cardiac surgery
3. patient with or at risk of cardiac arrhythmias
4. patients post cardiac arrest
5. patient with refractory status epilepticus
6. children with a greater than 5% leak around the endotracheal tube
7. children with a fraction of inspired oxygen >0.6

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critically ill children admitted on the intensive care unit at risk of developing fever
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Peters, MBBCh PhD, Principal Investigator — UCL Great Ormond Street Institute of Child Health

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Critically Ill Children With or Likely to Have Fever: Children above 10kg admitted to the paediatric intensive care unit at Great Ormond Street Hospital who are mechanically ventilated and have a high likelihood of developing a fever. Energy expenditure will be measured using indirect calorimetry at baseline, and continuously during fever, until fever subsides.
  Indirect calorimetry: Indirect calorimetry measurement at baseline (stable state), at onset of fever and continued till fever dehiscence
Period: Overall Study
Arm/Group | Critically Ill Children With or Likely to Have Fever
Started | 12
Completed | 3
Not Completed | 9
Not completed — Protocol Violation | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Febrile Critically Ill Children
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.7 [1.9 to 11.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12
Weight [Median (Inter-Quartile Range); unit: kilograms] | 16.9 [13.4 to 30.3]
Height [Median (Inter-Quartile Range); unit: centimetres] | 106 [86.5 to 140.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Energy Expenditure Per Degree Celsius During Fever and Defervescence
Description: Children at risk of fever will have energy expenditure measured by indirect calorimetry at baseline, when the develop a fever, and continuously until fever dehisces. Change in energy expenditure during fever to be calculated as difference in energy expenditure at the maximum temperature minus the energy expenditure at baseline, divided by the difference in temperature. Change in energy expenditure during defervescence to be calculated as difference in energy expenditure at the maximum temperature and the lowest temperature following the fall in temperature, divided by the difference in temperature.
  Both will also be expressed as a % of the starting energy expenditure (i.e. from baseline for change during fever, from maximum temperature during defervescence)
Time Frame: 6 hours
Population: Only one patient had a calorimetry measurement at baseline followed by a measurement during fever and two patients had measurements during fever, followed by fall in temperature.
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Change in Energy Expenditure During Fever: Children who had rise in temperature during Calorimetry measurement
- Change in Energy Expenditure During Fever Defervescence: Children who had a fall in temperature from a fever grade temperature (>=38C) during calorimetry
Arm/Group | Change in Energy Expenditure During Fever | Change in Energy Expenditure During Fever Defervescence
Number analyzed (Participants) | 3 | 2
percentage change | 18.8 (6.8) | 6.3 (6.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected till discharge from the paediatric intensive care unit. Typically this was 7 days
Groups:
- Critically Ill Children With or Likely to Have Fever: All Critically ill children with or likely to have fever who had calorimetry measurement
Arm/Group | Critically Ill Children With or Likely to Have Fever
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Only one patient had a calorimetry measurement at baseline followed by a measurement during fever and two patients had measurements during fever and defervescence thereafter. The hypothesis that energy expenditure increases by 10% from baseline during fever could not be accurately tested.

Recruitment was difficult because fever in ICU occurs early in admission when patients at their least stable enough for calorimetry. When stabilised, fever becomes less likely despite prior history.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT02939781/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT02939781/ICF_001.pdf